CLINICAL TRIAL: NCT07212738
Title: Post-stroke REhabilitation Start Evaluation for Reducing Vascular Events (PRESERVE)
Brief Title: Post-stroke REhabilitation Start Evaluation for Reducing Vascular Events
Acronym: PRESERVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Mohammed A Almekhlafi, MD, MSc, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB25-0152; 10040548 (Other Grant/Funding Number: UCalgary Research Excellence Chair)
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Ischemic Stroke
Keywords: stroke; rehabilitation; neuroimaging
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups after admission to hospital:
  1. Delayed care (group 1): active therapy beginning ≥3 days from symptom onset.
  2. Standard care (group 2): allied health assessment by 48 hours post-stroke followed by initiation of therapy at routine intensity (approximately 20 minutes/day of occupational and 20 minutes/day of physiotherapy). Therapy will depend on the level of disability of the participant, but will include working on standing, stepping, walking, balancing, self-care (i.e., grooming, dressing), functional task training (i.e., self-feeding), and addressing any cognitive and/or perceptive deficits.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be assigned to the control or experimental group using a 1:1 computer-generated randomized dynamic allocation procedure. All members of the research team will be blinded to group allocation. Participants and allied health team members (physiotherapist, occupational therapist, nursing) will not be blinded but will be asked not to tell the assessor or other participants which group they have been allocated to, in order to preserve blinding of the assessments. The study statistician and the rest of the Data Safety Monitoring Board will have access to the assignment if necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed mobilization (DeM) (Experimental): Active therapy beginning ≥3 days from stroke symptom onset.
  Interventions: Other: Delayed mobilization (DeM)
- Standard care (Active Comparator): Allied health assessment by 48 hours post-stroke followed by initiation of therapy at routine intensity (approximately 20 minutes/day of occupational and 20 minutes/day of physiotherapy). Therapy will depend on the level of disability of the participant, but will include working on standing, stepping, walking, balancing, self-care (i.e., grooming, dressing), functional task training (i.e., self-feeding), and addressing any cognitive and/or perceptive deficits.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Other: Delayed mobilization (DeM) — Delayed mobilization (group 1): active therapy beginning ≥3 days from symptom onset.
  Other Names: Standard care
  Arms: Delayed mobilization (DeM)
Other: Standard Care (in control arm) — Standard care (group 2): allied health assessment by 48 hours post-stroke followed by initiation of therapy at routine intensity (approximately 20 minutes/day of occupational and 20 minutes/day of physiotherapy). Therapy will depend on the level of disability of the participant, but will include working on standing, stepping, walking, balancing, self-care (i.e., grooming, dressing), functional task training (i.e., self-feeding), and addressing any cognitive and/or perceptive deficits.
  Active therapy will be conducted by the Foothills Medical Centre stroke unit (Calgary, AB, Canada) certified physiotherapists and occupational therapists. The allied health team will not be blinded to the randomization of participants.
  Arms: Standard care

SUMMARY:
The purpose of this research study is to better understand when to start rehabilitation therapies after acute ischemic stroke to prevent further harm to the brain and to improve outcomes for stroke survivors.

Stroke is the second leading cause of death and reduced quality of life worldwide, with one Canadian diagnosed with stroke every five minutes. The most common subtype, ischemic stroke, occurs when a blood vessel in the brain is blocked. Hyperacute treatments aim to remove these blockages to restore blood flow and improve deficits, but in some cases, this is not achieved and leads to persistent large or medium intracranial vessel occlusion.

After stroke, early medical and physical care can reduce physical and cognitive impairment and improve long-term functional outcomes. Prolonged immobilization can cause secondary complications and make recovery more difficult. Other research studies have demonstrated varying results with both benefit and no difference in the long-term level of functional independence when starting physical activity between 24 to 48 hours after acute ischemic stroke. The optimal timing for mobilization is unclear especially for patients with persistent vessel occlusion large stroke size, or intracranial hemorrhage, where starting active therapy too soon can cause additional harm by damaging the brain further.

In this research study, the investigators aim to evaluate the feasibility and effect of delayed mobilization (DeM), defined as physical therapy starting on or after day 3 from stroke symptom onset, on stroke volume growth and functional outcomes in patients with persistent vessel occlusion. The investigators think that individuals who still have evidence of persistent blockage in their arteries may benefit from waiting until day 3 after stroke to begin rehabilitation.

Improving care strategies for stroke survivors will ultimately benefit individuals, their families, and healthcare systems. This study may guide the optimal timing of initiating stroke rehabilitation in patients with persistent vessel occlusion and ischemia to improve recovery times and reduce long-term disabilities.

DETAILED DESCRIPTION:
While stroke remains the world's second leading cause of death and reduced quality of life in adults, mortality and disability have decreased over the years with advances in acute care and improvements in risk stratification (1). Ischemic stroke is the most common stroke subtype, caused by a blockage of blood flow in an artery in the brain. Revascularization interventions aiming to restore blood flow include intravenous thrombolysis and endovascular thrombectomy and have evidence in reducing the likelihood of long-term disability when performed rapidly in patients presenting early and without contraindications (2-4). Traditionally, functional independence is measured at 90 days after stroke using the modified Rankin scale (mRS) (5), where a score of 0 to 2 indicates limited impairment.

Early multidisciplinary care is essential for reducing physical and cognitive impairment following stroke, and in improving the chances of functional independence in the long-term. Immobilization for prolonged periods of time can result in secondary complications that further negatively impact recovery, including pneumonia, deep venous thrombosis, delirium, reduced muscle mass, and joint contractures (6). These secondary complications not only limit recovery, but increase the risk of mortality after stroke. Physical rehabilitation after stroke includes sitting, standing, supported ambulation, and repetitive body strength training with registered physiotherapists and occupational therapists. Early mobilization after stroke has been defined as starting physical rehabilitation between 24 to 48 hours after stroke onset, while some have proposed that very early (7) mobilization occurring within 12 hours of stroke onset has benefit.

Evidence for early or very early mobilization suggest that proteins associated with endogenous neural repair and growth-promoting factors are altered within the first few weeks after ischemic stroke (8-10). As a result, the upregulation in these processes may provide greater neuroplasticity for the injured brain to greater enhance its responsiveness to rehabilitation (11-13), and subsequently improve outcomes for stroke survivors. However, animal studies have also observed that starting exercise 6 hours after infarction raises pro-inflammatory cytokines and pro-apoptotic proteins leading to aggravated brain injury (14-15). The best timing for mobilization remains unclear when considering individual stroke factors such as persistent vessel occlusion (PVO), size of the ischemic core, or presence of intracranial hemorrhage, where active therapy can cause harm by increasing ischemic depolarization and reducing cerebral blood flow.

Clinically, the evidence regarding the timing of mobilization is additionally controversial. Studies have demonstrated both benefit (7,11,16-17) and no difference (18-22) in the level of functional independence following early mobilization between 24 to 48 hours after acute stroke when compared to individuals who received active therapy starting at 72 to 96 hours after stroke onset. More recently, the AVERT trial found a decrease in the odds of good outcomes (mRS score 0-2) at 3 months when mobilizing survivors within 24 hours of acute ischemic stroke (21). These findings are likely explained by their heterogenous sample including patients with PVO of large or medium caliber. Despite advances in stroke care and prevention, determining the optimal time to start physical activity after stroke to balance the risks of increasing stroke growth versus providing stroke survivors the best chance for greater independence is unknown.

Rehabilitation is crucial for reducing post-stroke disability and improving functional independence (23). The exact timing, however, on when to initiate rehabilitation after stroke is unclear. In some cases, starting rehabilitation immediately and very early after stroke (i.e., within 24 hours) can result in growth of the infarcted brain tissue due to cerebral hypoperfusion, resulting in worse clinical outcomes (21). In the present study, the investigators aim to determine the optimal timing of when to start active therapy after ischemic stroke by comparing a model of delayed mobilization (active therapy starting on or after day 3 post-stroke) to standardize care (active therapy starting by day 2 post-stroke). The investigators aim to determine the impacts of delayed mobilization on stroke volume growth, secondary brain injuries including hemorrhagic transformation and tissue hypoperfusion, and clinical measures of independence.

References

1. Donkor ES. Stroke in the 21st century: a snapshot of the burden, epidemiology, and quality of life. Stroke Res Treat. Nov 27, 2018;2018:3238165. doi:10.1155/2018/ 3238165.
2. Boulanger J, Lindsay M, Gubitz G, et al; Canadian stroke best practice recommendations for acute stroke management: prehospital, emergency department, and acute inpatient stroke care, update 2018. International Journal of Stroke. 2018;13(9):949-984.
3. Powers WJ, Rabinstein AA, Ackerson T, et al; Guidelines for the early management of patients with acute ischemic stroke: 2019 update to the 2018 guidelines for the early management of acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2019;50(12):e344-e418.
4. National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. New England Journal of Medicine. 1995;333(24):1581-1588.
5. Quinn TJ, Dawson J, Walters MR, Less KR. Functional outcome measures in contemporary stroke trials. Int J Stroke. 2009;4:200-206.
6. Bamford J, Dennis M, Sandercock P, Burn J, Warlow C. The frequency, causes and timing of death within 30 days of a first stroke: the Oxfordshire community stroke project. J Neurol Neurosurg Psychiatry. 1990;53(10):824-829.
7. Yanase L, Clark D, Baraban E, Stuchiner T. A Retrospective Analysis of Ischemic Stroke Patients Supports That Very Early Mobilization Within 24 Hours After Intravenous Alteplase Is Safe and Possibly Beneficial. J Neurosci Nurs. 2023 Dec 1;55(6):188-193.
8. Stroemer RP, Kent TA, Hulsebosch CE. Neocortical neural sprouting, synaptogenesis, and behavioral recovery after neocortical infarction in rats. Stroke. 1995;26:2135-2144.
9. Kawamata T, Alexis NE, Dietrich WD, Finklestein SP. Intracisternal basic fibroblast growth factor enhances behavioral recovery following focal cerebral infarction in the rat. J Cereb Blood Flow Metab. 1996;16:542-547.
10. Dahlqvist P, Zhao L, Johansson IM, Mattsson B, Johansson BB. Environmental enrichment alters nerve growth factor-induced gene A and glucocorticoid receptor messenger RNA expression after middle cerebral artery occlusion in rats. Neuroscience. 1999;93:527-535.
11. Biernaskie J, Chernenko G, Corbett D. Efficacy of rehabilitative experience declines with time after focal ischemic brain injury. J Neurosci. 2004 Feb 4;24(5):1245-54.
12. Dimyan MA, Cohen LG. Neuroplasticity in the context of motor rehabilitation after stroke. Nat Rev Neurol. 2011;7(2):76-85.
13. Johansson BB. Brain plasticity and stroke rehabilitation. The Willis lecture. Stroke. 2000;31(1):223-230.
14. Li F, Pendy JT Jr, Ding JN, Peng C, Li X, Shen J, Wang S, Geng X. Exercise rehabilitation immediately following ischemic stroke exacerbates inflammatory injury. Neurol Res. 2017;39(6):530-537.
15. Shen J, Huber M, Zhao EY, Peng C, Li F, Li X, Geng X, Ding Y. Early rehabilitation aggravates brain damage after stroke via enhanced activation of nicotinamide adenine dinucleotide phosphate oxidase (NOX). Brain Res. 2016;1648:266-276.
16. Wang F, Zhang S, Zhou F, Zhao M, Zhao H. Early physical rehabilitation therapy between 24 and 48 h following acute ischemic stroke onset: a randomized controlled trial. Disabil Rehabil. 2022;44(15):3967-3972.
17. Langhorne P, Stott D, Knight A, Bernhardt J, Barer D, Watkins C. Very early rehabilitation or intensive telemetry after stroke: a pilot randomised trial. Cerebrovasc Dis. 2010;29(4):352-360.
18. Anjos JM, Neto MG, de Araújo Tapparelli Y, Tse G, Biondi-Zoccai G, de Souza Lima Bitar Y, Roever L, Duraes AR. Efficacy and safety of very early mobilization after thrombolysis in acute ischemic stroke: a randomized clinical trial. J Neurol. 2023 Feb;270(2):843-850.
19. Sundseth A, Thommessen B, Ronning OM. Early mobilization after acute stroke. J Stroke Cerebrovasc Dis. 2014;23(3):496-499.
20. Sundseth A, Thommessen B, Ronning OM. Outcome after mobilization within 24 hours of acute stroke: a randomized controlled trial. Stroke. 2012;43(9):2389-2394.
21. AVERT Trial Collaboration group. Efficacy and safety of very early mobilisation within 24 h of stroke onset (AVERT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):46-55.
22. Bernhardt J, Dewey H, Thrift A, Collier J, Donnan G. A Very Early Rehabilitation Trial for Stroke (AVERT): phase II safety and feasibility. Stroke. 2008;39:390-396.
23. Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, et al. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014;9(2):e87987.

ELIGIBILITY:
Inclusion Criteria:

* Participants with acute ischemic stroke presenting to Foothills Medical Centre meeting eligibility for intravenous thrombolysis (Tenecteplase, TNK) - ≥18 years of age presenting within 4.5 hours of symptom onset with a diagnosis of suspected acute ischemic stroke causing significant neurological disability - and/or endovascular thrombectomy (EVT).
* Age ≥18 years.
* Persistent vessel occlusion will be defined as any of the following:

  * EVT treatment of medium or large intracranial vessel occlusion with a thrombolysis in cerebral infarction (TICI) score of ≤2b.
  * A moderate infarct core (ASPECTS ≤5) despite TICI 3.
  * 24-hour CT with evidence of hyperdense sign appropriate to clinical deficits.

Exclusion Criteria:

* Comorbid conditions limiting recovery or life expectancy (e.g., significant cognitive impairment, stage IV cancer, end-stage renal disease).
* Low pre-stroke baseline functional status (mRS ≥4).
* Symptoms due to another acute neurological condition (e.g., migraine with aura, seizure) or neurological deficits secondary to metabolic/toxic derangements (e.g., hyponatremia, hypoglycemia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of delayed mobilization. | Participants will be assessed for up to 3 months post-stroke, predominantly on their 7 day admission and at their 3-month outpatient follow-up (8 total days).
  Our primary outcome will be completion of the trial to determine whether delaying mobilization is feasible.

SECONDARY OUTCOMES:
Incidence of secondary neurovascular injury. | Neuroimaging outcomes will be compared from admission (day 1-2 post-stroke) to repeat MRI on day 7.
  The secondary objective is to determine the incidence of secondary neurovascular injury (i.e., infarct growth and/or hemorrhagic transformation) in individuals with delayed mobilization. MRI brain scans at 1-2 day after admission to hospital and on day 7 after stroke will be used to measure stroke volume growth following intervention, comparing the metrics to the baseline scans.

OTHER OUTCOMES:
Rate of functional independence. | Participants will be assessed for up to 3 months post-stroke, predominantly on their 7 day admission and at their 3-month outpatient follow-up (8 total days).
  The tertiary objective is to assess if delayed mobilization is associated with greater rehabilitation candidacy and improved functional outcomes (modified Rankin scale [mRS] score of 0-2) at 3 months. The scores from hospital discharge and at 3-month follow-up will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No